CLINICAL TRIAL: NCT04209153
Title: Evaluation of the Effect of Transcranial Direct Current Stimulation (tDCS) in Nicotine-Dependent Tobacco Users
Brief Title: Direct Transcranial Electrical Stimulation in Tobacco Addiction (tDCS)
Acronym: tDCS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190731; 2019-A01946-51 (Other: IDRCB)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Adults (Male and Female Subjects) With Tobacco Dependence
Keywords: Tobacco; addiction; transcranial non invasive direct brain stimulation; adults
MeSH Terms: conditions — Behavior, Addictive | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — tDCS sessions (with Direct Transcranial Electrical Stimulation (tDCS) device - Neuroelectrics

SUMMARY:
In summary, there are currently many therapeutic tools for achieving some degree of control or even cessation of tobacco addictive use. No single therapy seems to have proven itself sufficiently effective to be the preferred treatment axis in the management of this addiction. We can also point out that so far the main treatments aimed at reducing or controlling the craving phenomenon are of a pharmacological nature, thus exposing the participants to the side effects inherent to this type of treatment. In this perspective, the establishment of non invasive brain stimulation (TdCS), acting in a targeted manner on craving and whose effects would be mild and transient, appears quite justified, especially in addition to psychotherapy. In the context of the management of addictive pathologies, the choice of smoking dependence seems relevant to us insofar as this addiction represents a major public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* Nicotine dependent subjects according to the Fagerström test (score ≥5)
* Subjects consuming daily tobacco.
* Subjects understanding and reading French and able to express themselves in this language.
* Signed informed consent to participate indicating that the subject has understood the purpose and the procedures required by the study and agrees to participate in the study and to comply with the requirements and limitations of this study
* Affiliation to the French social security scheme or beneficiary of such a scheme.
* No other method to decrease or stop smoking at the same time as the study.

Exclusion Criteria:

* Guardianship
* Pregnant or lactating woman
* Patient under AME
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File".
* Subjects with intracranial hypertension
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator.
* Treatment with buproprion or varenicline in progress
* Episode or family history of epilepsy, convulsion.
* Disease causing damage to the brain (aneurysm, tumor, ...).
* Cochlear or ocular implant.
* Stimulator or cardiac defibrillator.
* Presence of metal in the skull (clip on aneurysm, prosthesis, ...).
* Eczema on the scalp.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All tobacco smokers who will ask for consultation in our ward.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-05-29 (Estimated)

PRIMARY OUTCOMES:
Fagerström score (3 is the highest score and O the lowest one for item 1. A score of 1 or 2 means low dependence (for item 1 only as well as if you use the total score) | 15 days
  average difference in Fagerström score 1 scores that assess craving for tobacco between pre-treatment assessment (J0) and short-term post-treatment evaluations (J15).

SECONDARY OUTCOMES:
tobacco consumption | 15 days
  Evaluation of changes in tobacco consumption and smoking craving intensity and tolerance of tDCS

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrie Adultes Et Addictologie, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No